CLINICAL TRIAL: NCT02100215
Title: Quantifying the Influence of Expert Modeling on Novice Nurse Competence and Self-Efficacy
Brief Title: Quantifying the Influence of Expert Modeling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Ashley Franklin, Instructor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MPtSim-Ashland
Record Dates: First submitted 2014-03-24; First posted 2014-03-31 (Estimated); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Competence; Self-efficacy
Keywords: simulation; competence; self-efficacy; novice nurses

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Expert Modeling (Experimental): Participants will have access to 70 minutes of expert modeling videos available over 5 weeks on an online learning management system. The investigator will be the expert model in the videos. Expert modeling videos will address content related to seven concepts: Taking report with a graphic organizer worksheet, prioritizing patient care, delegating to unlicensed assistive personnel, safety checks in patient rooms, focused physical assessments, safe medication administration, and using a standardized healthcare provider communication tool on the telephone.
  Interventions: Other: Common readings and educational handouts; Other: Expert Modeling
- Voice Over PowerPoint (Active Comparator): Participants will have access to 60 minutes of voice over PowerPoint slides, available over 5 weeks on an online learning management system, specifically to match exposure and content with the expert modeling video group. The script for PowerPoint will contain content related to the aforementioned seven concepts. There will be static photos, but no expert modeling videos, on PowerPoint slides. The investigator will narrate the voice over PowerPoint.
  Interventions: Other: Common readings and educational handouts; Other: Voice Over Power Point
- Reading (Placebo Comparator): Participants will have access to articles, policies, and procedures on an online learning management system. The estimated time required for participants to review these materials is 45 minutes
  Interventions: Other: Common readings and educational handouts

INTERVENTIONS:
Other: Common readings and educational handouts — Participants in all groups have common readings related to policies for nursing care in acute care facilities. There will be additional handouts related to performing safety checks and a focused physical assessment.
Other: Expert Modeling — 70 minutes of expert modeling videos
  Arms: Expert Modeling
Other: Voice Over Power Point — 60 minutes of Voice Over PowerPoint presentations
  Arms: Voice Over PowerPoint

SUMMARY:
The purpose of this study is to learn more about the effects of various types of simulation preparation methods on novice nurses' competence and self-efficacy. Participants will be recruited from an academic course (N424 Integrated Practicum). Participants will be randomized to three intervention groups (i.e. expert modeling video, voice over PowerPoint, and traditional readings). All participants will complete self-efficacy surveys and two simulations. During simulation, participants will be scored based on their competence according to a performance rubric. The hypothesis is that participants in the expert modeling group will demonstrate more change in competence and report more change in self-efficacy scores than participants in other groups.

DETAILED DESCRIPTION:
Investigators will compare self-confidence and competence scores between the three groups after the pre-test and posttest simulations. The self-efficacy survey is an 7-item scale that involves participants rating their self-efficacy about providing care for multiple patients. Participants rate their self-efficacy on a 1 to 5 (not confident to very confident scale). The survey takes 5 minutes to complete. The self-efficacy survey has been used in many simulation research studies previously with novice nurses. Competence will be measured with a rater-observation measure which has previously been used in simulation research.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in capstone clinical course
* Oregon Consortium for Nursing Education curriculum
* Ashland, OR

Exclusion Criteria:

* No exclusion criteria

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Creighton Simulation Evaluation Instrument | Change from baseline on Creighton Simulation Evaluation Instrument at 5 weeks

SECONDARY OUTCOMES:
National League for Nursing Student Satisfaction and Self-Confidence with Learning scale | Change from baseline on NLN Student Satisfaction and Self-Confidence with Learning scale at 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Franklin, Principal Investigator — Oregon Health and Science University; Christopher S Lee, PhD, Study Chair — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, School of Nursing, Ashland, Oregon, United States